CLINICAL TRIAL: NCT01091675
Title: Assessment of the Response to Etoricoxib in Patients With Ankylosing Spondylitis (AS) and Inadequate Response to ≥2 Nonsteroidal Antiinflammatory Drug (NSAID)
Brief Title: Assessment of the Response to Etoricoxib in Patients With Ankylosing Spondylitis and Inadequate Response to ≥2 NSAIDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Foundation of Rheumatology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRE-2009-01; 2009-017309-12 (EudraCT Number)
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; biologic therapies; ASAS; ASASBIO; etoricoxib; NSAIDs; COX-2 Inhibitor; ARCOXIA 90 mg; BASDAI Bath Ankylosing Spondylitis Disease Activity Index
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etoricoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- etoricoxib (Experimental): All the patients who fulfil the eligibility criteria will start a 4-week open label treatment period to evaluate the response to treatment with etoricoxib 90 mg.
  Interventions: Drug: Etoricoxib

INTERVENTIONS:
Drug: Etoricoxib — Etoricoxib 90 mg/day/PO during 4 weeks Positive response to the therapy (in investigator opinion): Ongoing treatment with 90 mg/day/PO until 24 weeks.
  Other Names: Arcoxia

SUMMARY:
The goal of this research is to assess the percentage of non-responders to ≥ 2 NSAIDs candidates a biological therapy that could adequately respond to treatment with etoricoxib This study confirm the result of a previous study in a wider similar population. Basing on previous results, the response rate will be assessed by ASASBIO criteria. The efficacy of the treatment with etoricoxib 90 mg will be assessed at week 4 in a population of patients with AS who didn't respond adequately to a previous therapy with ≥ 2 NSAIDs.

Those patients that, based on the ASABIO criteria, achieved a sufficient clinical response will be followed until week 24 to asses the maintenance of the study drug effects.

DETAILED DESCRIPTION:
Etoricoxib is an oral, selective cyclooxygenase 2 inhibitor approved for the symptomatic treatment of ankylosing spondylitis (AS) in Spain.

Etoricoxib is a marketed product indicated for the relief of symptomatic osteoarthritis, rheumatoid arthritis, ankylosing spondylitis, pain and signs of inflammation associated with acute gouty arthritis. In ankylosing spondylitis,the recommended dose is 90 mg once daily.

Clinical pharmacology studies demonstrate that Etoricoxib induce dose-dependent inhibition of COX-2 without inhibit COX-1, up to 150 mg daily dose.

Etoricoxib did not inhibit the gastric synthesis of prostaglandin and had no effect on platelet function. Cyclooxygenase is responsible for the prostaglandin synthesis. Were identified two different isoforms of cyclooxygenase, COX-1 and COX-2. It has been shown that COX-2 is the major enzyme responsible for the synthesis of prostanoid mediators involved in pain, inflammation and fever.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years.
2. Patients with diagnosis of AS (based on New York criteria) made ≥ 6 months prior to study start.
3. Patient with axial involvement.
4. Patients who have been treated with ≥ 2 documented NSAID with proven anti-inflammatory potency during at least 3 months at maximal recommended or tolerated doses prior the visit 1.
5. Patients who demonstrate a Bath Ankylosing Spondylitis Disease Activity Index score of ≥ 4 (range 0-10).

Exclusion Criteria:

1. Patient that according to the investigator opinion is legally unable (i.e. mentally incapable person), with psychiatric disorder precedent, active psychosis or emotional problems at the moment to be enrolled in the study.
2. Patient who is participating in a clinical study with a drug or experimental device or it was done within 4 weeks prior to the inform consent signature.
3. Patient with a recent history (since last 5 years) of abuse or dependence to opiates, tranquilizer or drugs at the inform consent signature moment. Patient with a recent history (since last 5 years) of alcoholism or drug addiction.
4. Patient with a history of neoplastic disease or malignant neoplasia ≤ 5 years prior to the inform consent signature, except basal cell or squamous cell cancer skin adequately treated or uterine cancer insitu without recurrence prior to study entry according to the investigator opinion. Patients with history of leukemia, lymphoma, malignant melanoma or myeloproliferative disease cannot participate at the study.
5. Pregnancy, lactation or waiting to conceive a child
6. Patient with history of disorders, treatments or laboratory abnormality that can interfere with the study results and study participation.
7. Patient cannot comply with the study procedures, study calendar. Patient with plan of moving.
8. Patients awaiting the legal assessment of the degree of disability or the permanent work disability
9. Patients unable to respond to questionnaires (difficulty understanding and / or reading of questionnaires)
10. Any other warning that, in the investigator opinion, could discourage the inclusion of the patient in the study.
11. Patient to be treated with other drug which can modulate the pain perception
12. Patients with AS associated disease (inflammatory bowel disease, psoriasis).
13. Patients with active peripheral articular involvement defined by presence of peripheral arthritis.
14. Patient with predominant enthesitis or an enthesis that, according to investigator's opinion, can confound the correct evaluation.
15. Presence of extra-articular manifestations.
16. Patients with fibromyalgia or other rheumatic disorders that could confound the evaluation of efficacy
17. Patients with AS who received biologic therapy. Note: The use of approved nonstudy antirheumatic therapy at a stable dose(methotrexate, sulfasalazine) for 3 months prior to the study start will be allowed.
18. Patients with AS who received active treatment with etoricoxib
19. Hypersensitivity to the active substance or to any of the excipients
20. Active peptic ulceration or active gastro-intestinal bleeding
21. Patients with severe renal failure (creatinine clearance rate < 30 ml/min)
22. Congestive heart failure (NYHA II-IV)
23. Established ischaemic heart disease or cerebrovascular disease
24. Patients with severe hepatic dysfunction (serum albumin <25 g/l or Child-Pugh score ≥10).
25. Patients who have experienced bronchospasm, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria, or allergic-type reactions after taking acetylsalicylic acid or NSAIDs including cyclooxygenase-2 inhibitors
26. Patients with hypertension whose blood pressure is persistently elevated above 140/90mmHg and has not been adequately controlled

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Gratacós, PhD/ MD, Principal Investigator — Parc Tauli Hospital; Eduardo Collantes Estevez, PhD/ MD, Principal Investigator — Reina Sofia Hospital; Xavier Juanola Roura, PhD/MD, Principal Investigator — Bellvitge Hospital; Raimon Sanmartí Sala, PhD/MD, Principal Investigator — Hospital Clinic i Provincial Barcelona; Juan Mulero Mendoza, PhD/MD, Principal Investigator — Puerta de Hierro Hospital; Estefania Moreno Ruzafa, PhD/MD, Principal Investigator — San Rafael Hospital; Luis Francisco Linares Ferrando, PhD/MD, Principal Investigator — Virgen de la Arrixaca Hospital; Rubén Queiro Silva, PhD/MD, Principal Investigator — Asturias Hospital; Elia Brito Brito, PhD/MD, Principal Investigator — Ramon y Cajal Hospital; Carlos Alberto Montilla Morales, PhD/MD, Principal Investigator — Hospital Clinic of Salamanca; Maria Cruces Fernández Espartero, PhD/MD, Principal Investigator — General de Mostoles Hospital; Pilar Fernández Dapica, PhD/MD, Principal Investigator — University Hospital 12 de Octubre; Rosario García de Vicuña, PhD/MD, Principal Investigator — University Hospital de la Princesa; Rosa Morlá, PhD/MD, Principal Investigator — Sant Pau i Santa Tecla Hospital
Locations (14):
- Spain (14):
  - Sant Rafael Hospital, Barcelona, Barcelona
  - Clinic I Provincial Hospital, Barcelona, Barcelona
  - Bellvitge Hospital, Barcelona, Barcelona
  - Parc Tauli Hospital, Sabadell, Barcelona
  - Reina Sofia University Hospital, Córdoba, Cordoba
  - Ramon Y Cajal Hospital, Madrid, Madrid
  - University Hospital 12 Octubre, Madrid, Madrid
  - Puerta de Hierro Hospital, Madrid, Madrid
  - Hospital General of Mostoles, Madrid, Madrid
  - Virgen de la Arrixaca Hospital, Murcia, Murcia
  - Central Hospital of Asturias, Oviedo, Principality of Asturias
  - Hospital Clinic of Salamanca, Salamanca, Salamanca
  - University Hospital de la Princesa, Madrid
  - Sant Pau i Santa Tecla Hospital, Tarragona

REFERENCES:
- [Background] Estévez, E. Collantes, and A. Escudero Contreras.
- [Background] Sociedad Española de reumatología: estudio EPISER. Prevalencia de las enfermedades reumáticas en la población española. Reumatología. Madrid, Merck, Sharp & Dohme, 2001.
- [Background] van der Heijde D, Baraf HS, Ramos-Remus C, Calin A, Weaver AL, Schiff M, James M, Markind JE, Reicin AS, Melian A, Dougados M. Evaluation of the efficacy of etoricoxib in ankylosing spondylitis: results of a fifty-two-week, randomized, controlled study. Arthritis Rheum. 2005 Apr;52(4):1205-15. doi: 10.1002/art.20985. PMID 15818702
- [Background] Jarrett SJ, Sivera F, Cawkwell LS, Marzo-Ortega H, McGonagle D, Hensor E, Coates L, O'Connor PJ, Fraser A, Conaghan PG, Emery P. MRI and clinical findings in patients with ankylosing spondylitis eligible for anti-tumour necrosis factor therapy after a short course of etoricoxib. Ann Rheum Dis. 2009 Sep;68(9):1466-9. doi: 10.1136/ard.2008.092213. Epub 2008 Oct 24. PMID 18952641
- [Background] Braun J, Pham T, Sieper J, Davis J, van der Linden S, Dougados M, van der Heijde D; ASAS Working Group. International ASAS consensus statement for the use of anti-tumour necrosis factor agents in patients with ankylosing spondylitis. Ann Rheum Dis. 2003 Sep;62(9):817-24. doi: 10.1136/ard.62.9.817. PMID 12922952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 58 patients in total, with ankylosing spondylitis, and Inadequate response to ≥2 NSAIDs. Patients who met The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) scores of 4 or higher and all study criteria participate in the study and were randomized at 14 study sites. The last patient completed in May 2013.
Pre-assignment Details: From a total of 58 patients recruited 1 did not met the exclusion criteria, so 57 patients start the first phase. 4 patients abandoned the study due to hypertension. 53 patients completed the first phase. 27 did not proceed to phase 2 due to lack of efficacy and 3 patients were withdraw due to hypertension. 23 patients complete the study period.
Period: Overall Study
Arm/Group | Etoricoxib
Started | 57 (7 patients leave the study due to hypertension, 27 patients withdrew due to lack of efficacy)
Completed | 23
Not Completed | 34
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 27

BASELINE CHARACTERISTICS:
Arm/Group | Etoricoxib
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] — From a total of 58 patients recruited one did not met the exclusion criteria so 57 patients were included in the study.
  years | 44 [23 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 58

OUTCOME MEASURES:

1. Primary Outcome: the Percentage of Patients Fulfilling the Assessment Study (ASAS) Response Criteria Were Determined
Description: BASDAI Bath Ankylosing Spondylitis Disease Activity Index, is the gold standard for measuring and evaluating disease activity in Ankylosing Spondylitis consists of a one through 10 scale which is used to answer 6 questions pertaining to the 5 major symptoms of AS.
  BASDAI has been used to assess the efficacy of the treatment. Possible Patients were considerate respond to ASABIO criteria when presented a change of 2 in the BASDAI score range.
Time Frame: the ASAS response were evaluated at week 2 and 4 and after 6 months treatment
Population: Patients with physician-diagnosed Ankylosing Spondylitis at 6 months before study start
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etoricoxib
Number analyzed (Participants) | 57
percentage of participants | 19 [10 to 30]

ADVERSE EVENTS:
Time Frame: from September 23rd 2010 until May 28th 2013
Arm/Group | Etoricoxib
Serious Adverse Events (participants affected / at risk) | 1/57
Other Adverse Events (participants affected / at risk) | 20/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib (N=57)
cavernous hemangioma (Vascular disorders) | 1 (1) — The investigator evaluated this serious adverse event SAE, as possibly related to the study drug, The patient already suffered from cavernoma pedunculi left quadrigeminy but was unknown until symptoms appearance. Was withdrawn from the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etoricoxib (N=57)
arterial hypertension (General disorders) | 7 — 7 patients were withdrew from the study due to hypertension. 1 case certainly related to the study drug. 3 patients demonstrate seriousness grade 1, and grade 2 in 4 patients
Tachycardia (Cardiac disorders) | 3
headache (Nervous system disorders) | 2
anxiety (General disorders) | 2
Nervousness (General disorders) | 2
cold (General disorders) | 2
upper respiratory infection (Infections and infestations) | 1
weight gain (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other